CLINICAL TRIAL: NCT00459589
Title: Nutritional Intervention in Geriatric Oncology in Patients at Risk of Undernutrition
Brief Title: Nutritional Intervention in Geriatric Oncology
Acronym: INOGAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Ministry of Health, France (Other Government); Ligue contre le cancer, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CHUBX 2006/11; 2006/018
Record Dates: First submitted 2007-04-11; First posted 2007-04-12 (Estimated); Last update posted 2012-06-20 (Estimated); Status verified 2012-06

CONDITIONS: Cancer; Undernutrition; Aging
Keywords: Cancer; elderly; malnutrition; chemotherapy; survival; comprehensive geriatric assessment; morbidity
MeSH Terms: conditions — Neoplasms; Malnutrition | interventions — Nutritionists

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): nutritional intervention with dietician at each cycle of chemotherapy in 6 first cycles to maintain 30 kcal/kg/d and 1.2 protein/kg/d
  Interventions: Behavioral: nutritional intervention with dietician plus usual nutritional care
- 2 (Active Comparator)
  Interventions: Behavioral: usual nutritional care

INTERVENTIONS:
Behavioral: nutritional intervention with dietician plus usual nutritional care — nutritional intervention with dietician at each cycle of chemotherapy in 6 first cycles to maintain 30 kcal/kg/d and 1.2 protein/kg/d
  Arms: 1
Behavioral: usual nutritional care — usual nutritional care
  Arms: 2

SUMMARY:
Older patients with cancer are poorly treated or not treated at all. A previous study in the south west of France (364 patients) showed that patients receiving chemotherapy had short survival times which strongly depended on nutritional status. In this study, the researchers would like to evaluate if individual dietician follow-up at each cycle of chemotherapy increases survival of patients at risk of undernutrition.

DETAILED DESCRIPTION:
Undernutrition in patients with cancer also called tumour cachexia concerns about 50% of this population during tumour progression. It's well established that loss of weight is poor prognosis factor in patients treated by chemotherapy in digestive cancers. Small number of studies assessing undernutrition, its management and consequences on prognosis were published. Previous study lead by our team in oncogeriatry in Aquitaine accrued 364 patients more than 70 years old and treated by chemotherapy for cancer. Median follow-up at 13 months for intermediary analysis about 155 first patients revealed at first geriatric evaluation, 28 pts (18.7%) were malnourished (MNA<17) and 72 pts (48.0%) at risk of malnutrition (MNA 17 to 23.5). At one year median follow-up major mortality was observed in 20 (71.4%) undernourished patients, 34 (47.2%) patients at risk of undernutrition and 13 (26.0%) patients without nutritional problem. According to consensus undernourished patients received nutritional support. Management of patients at risk of malnutrition is not clear. Our hypothesis is that nutritional support in patients at risk of undernutrition detected during geriatric evaluation could increase survival, safety, functional status and quality of life of patients. We construct an open multicentric two group randomized trial comparing usual nutritional management versus usual nutritional management plus nutritional intervention with dietician at each cycle of chemotherapy in 6 first cycles to maintain 30 kcal/kg/d and 1.2 protein/kg/d. Principal objective is to increase survival at 1 year with 10%. According to O'Brien and Fleming method we have to include 410 pts in each group, about 1640 pts will be evaluated by MNA test.

ELIGIBILITY:
Inclusion Criteria:

* Over 70 years of age
* Histologically proven cancer
* Treatment by chemotherapy
* Risk of undernutrition according to MNA score between 17 and 23.5
* ECOG ≤ 3
* Life expectancy > 12 weeks
* Patient affiliated with the French social security regimen
* Written informed consent

Exclusion Criteria:

* MNA score under 17 or over 23.5
* Geographic, psychological, or social conditions potentially hampering compliance with the study protocol
* Symptomatic central nervous system (CNS) metastases
* Chemotherapy treatments not published as standard protocols
* Treatment that does not allow geriatric evaluation and dietician follow-up.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 341 (Actual)
Dates: Start 2007-04; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Survival | 1 year

SECONDARY OUTCOMES:
Survival | 2 years
toxicity of chemotherapy (NTC CTCv3 scale) | within 6 cycles of chemotherapy treatment,
quality of life | before and after chemotherapy treatment
biology (C-reactive protein [CRP], albumin, haemoglobin, creatinine clearance) | before and after treatment
mood (GDS-15) | before and after treatment
function: IADL, ADL, get up and go test | before and after treatment
weight | before and after treatment
MNA | before and after treatment
dietary intakes | before and after treatment
hospitalisation frequency | during treatment
opportunistic infection frequency | during treatment
fall, breaks, pressure sore | during treatment
death | during treatment and at 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle BOURDEL MARCHASSON, Pr., Principal Investigator — University Hospital, Bordeaux, France; Geneviève CHENE, Pr., Study Chair — University Hospital, Bordeaux, France
Locations (2):
- France (2):
  - Institut Bergonié - 229 Cours de l'Argonne, Bordeaux
  - Pôle de Gériatrie - CHU Bordeaux-Hôpital Xavier Arnozan - Avenue du Haut-Lévèque, Pessac

REFERENCES:
- [Derived] Bourdel-Marchasson I, Blanc-Bisson C, Doussau A, Germain C, Blanc JF, Dauba J, Lahmar C, Terrebonne E, Lecaille C, Ceccaldi J, Cany L, Lavau-Denes S, Houede N, Chomy F, Durrieu J, Soubeyran P, Senesse P, Chene G, Fonck M. Nutritional advice in older patients at risk of malnutrition during treatment for chemotherapy: a two-year randomized controlled trial. PLoS One. 2014 Sep 29;9(9):e108687. doi: 10.1371/journal.pone.0108687. eCollection 2014. PMID 25265392